CLINICAL TRIAL: NCT07210853
Title: Postural Stability and Balance Impairments in Non-Athletic Individuals After Anterior Cruciate Ligament Reconstruction: A Cross-Sectional Study
Brief Title: Postural Stability Following Anterior Cruciate Ligament Reconstruction
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Gürkan Demirtas, PhD, Nigde Omer Halisdemir University
Other Study IDs: E-95860085-050.02.04-453062
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament (ACL); Postural Stability
Keywords: anterior cruciate ligament; balance; postural stability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACL: individuals with a history of ACL reconstruction
- Control: healthy controls matched to the ACL group

SUMMARY:
Anterior cruciate ligament (ACL) injuries are among the most frequent knee injuries, often leading to deficits in postural stability and balance as a result of mechanoreceptor damage, which disrupts proprioceptive feedback and sensorimotor regulation. The present study aimed to provide a detailed evaluation of postural stability and balance in non-athletic individuals following ACL reconstruction (ACLR).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-40 years who had undergone unilateral ACLR Tegner activity score of ≥ 5

Exclusion Criteria:

* Any other orthopedic conditions affecting the lower extremities besides ACL injury

A history of lower extremity surgery for any reason

Lower limb malalignment

Neurological or circulatory disorders that could impair balance

Visual or vestibular problems

Rheumatologic diseases

Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included 58 non-athletic individuals aged 18-40 years. Among them, 29 participants had undergone unilateral anterior cruciate ligament reconstruction (ACLR) 12-24 months prior to the study, and 29 healthy individuals matched for age, height, weight, and sex served as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Static Balance- Bipodal stance test | baseline
Static balance- Single-leg stance test | baseline
Dynamic Balance- Y-Balance Test | baseline

SECONDARY OUTCOMES:
KOOS (Knee Injury and Osteoarthritis Outcome Score) | baseline
IKDC (International Knee Documentation Committee - Subjective Form) | baseline
Tegner Activity Scale | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Niğde Ömer Halisdemir Üniversitesi, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No